CLINICAL TRIAL: NCT01819077
Title: Register Study: TMMR and Therapeutic Lymphadenectomy According to M.Hoeckel for Treatment of Cervical Cancer FIGO IB-IIA
Brief Title: TMMR (Total Mesometrial Resection) Register Study
Acronym: TMMR-RS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Dr. Paul Buderath, Prof. Dr. med. Rainer Kimmig, University Hospital, Essen
Other Study IDs: TMMR-RS
Record Dates: First submitted 2013-03-19; First posted 2013-03-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; TMMR; therapeutic lymphadenectomy; register study
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TMMR: Patients with cervical cancer Stages IB - IIA treated with TMMR and tLNE
  Interventions: Procedure: TMMR

INTERVENTIONS:
Procedure: TMMR — Radical hysterectomy by Total Mesometrial Resection (TMMR) and therapeutic lymphadenectomy (tLNE)

SUMMARY:
TMMR/tLNE was shown to result in very low locoregional recurrence rates and low morbidity in surgical treatment of cervical cancer stage IB-IIA without any adjuvant radiotherapy even in high risk situations. More and more this therapeutic strategy is implemented in clinical routine in specialized cancer centres, thus, treatment of cervical cancer could be performed for these stages in a systematically defined and reproducible radicality; adjuvant radiotherapy could be spared for recurrent disease, thus lowering morbidity and resource assignment in primary treatment dramatically. Due to the nerve-sparing character of the procedure bladder, bowel and sexual dysfunction would also be minimized and markedly benefit the patient.

This study is designed to follow up the results of this therapeutic concept adapted to clinical routine in a multiinstitutional register study accompanied by detailed assessment of pathological work-up, quality of life and bladder and sexual function following surgery.

DETAILED DESCRIPTION:
Rationale for the multimodal treatment of cervical cancer in FIGO stages IB-IIA according to M. Hoeckel: Total mesometrial resection (TMMR) is a newly developed procedure for surgical treatment of cervical cancer of FIGO stage IB to IIB. The procedure is based on embryologically determined surgical anatomy that was generated from investigations of the embryonal and fetal development of the Müllerian organ system and of local tumor spread of cervical cancer at the macroscopic, microscopic and molecular level (11-13). The observation that the cervical cancer follows the embryologically derived compartment hierarchy led to the definition of a new principle of radicality for oncological surgery, i.e., the resection of a tumor within the borders of the compartment representing the morphogenetic unit of the tumor origin. A resection that follows this principle leads to high local control (>95%) without additional radiotherapy. The resection line of the vagina is located inside the compartment, therefore intraoperative frozen section examination of the TMMR specimen is necessary to achieve wide margins. Adjacent structures that belong to another morphogenetic unit can be saved in spite of immediate proximity to the tumor. The autonomic nerves are saved with the TMMR concept as well as the ureters, the urinary bladder and their mesenteries containing all blood vessels, and the rectum with the mesorectum.

Therapeutic LNE: With TMMR tLNE has to be done with therapeutic intent, so that in case of lymph node metastases a high regional tumor control without adjuvant radiotherapy can be achieved (27). Therapeutic pelvic tLNE needs the removal of the lymph node groups within the scope of the classical systematic pelvic LNE and additionally, the paravisceral fatty tissue inferior to the obturator nerve, perispinal, gluteal and presacral lymph nodes to S2. The therapeutic pelvic LNE is done with exposition and protection of the plexus hypogastricus superior, the nervus hypogastricus and the plexus hypogastricus inferior and all ureter supplying vessels, bilaterally. In case of intraoperative evidence of pelvic lymph node metastases in first line nodes stepwise ascending therapeutic para-aortic LND with protection of the plexus hypogastricus superior and the nervi splanchnici lumbales has to be done. To date no prospective, randomized trial has proven a survival benefit of adjuvant chemotherapy alone in patients with early cervical cancer and histopathological risk factors. However, retrospective studies and the results of Peters et al. (20), comparing adjuvant chemo-radiotherapy with radiotherapy alone in patients after surgery for cervical cancer suggest that adjuvant chemotherapy may exert an impact on survival. The possible effect of adjuvant chemotherapy should be taken into consideration when applying only surgical therapeutic concepts (23;25). Therefore, adjuvant chemotherapy in case of risk factors was performed Hoeckel's trial. The mono-institutional prospective study of the University of Leipzig, Department of Gynecology and Obstetrics, has shown that the treatment concept for cervical cancer FIGO stages IB-IIB including TMMR and therapeutic LNE without adjuvant radiotherapy achieves a markedly improved therapeutic index in comparison with historic controls (16;22): locoregional control was 96% versus 91%, relapse-free survival after three years was 93% vs. 84%, treatment-caused side effects were 9% exclusively grade II vs. 28% grade II and III (11-13).

Scientific aims

1. Observation of results of standardization of radical hysterectomy and therapeutic lymphadenectomy in cervical cancer FIGO IB -IIA on the basis of ontogenetically defined compartment theory in a multicentric approach by TMMR/LND in clinical routine
2. Assessment of locoregional recurrence in this concept without any radiation therapy showing that postoperative irradiation and associated morbidity can also be avoided and irradiation may be maintained for rescue in recurrency under conditions of clinical routine
3. Confirmation of the low morbidity of TMMR due to autonomous nerve and vessel preservation by concomitant urogynecological and psychosexual subprotocols in clinical routine treatment

Requirements for participating centers of the register study

1. Study of educational video (M. Hoeckel, Leipzig 2010; R. Kimmig, Essen 2012)
2. Passed Participation of 2 day educational training concerning TMMR at "Leipzig School of Oncological Surgery"
3. Performing at least 10 TMMR procedures at participating institution/year
4. Evaluation of surgical technique at the participating institution by Prof. Hoeckel (Leipzig) or Prof. Kimmig (Essen) or substitute determined by M.Hoeckel or R. Kimmig
5. Securing standardized workup of the surgical specimen by pathologists according to the protocol (Prof. Horn, Leipzig)
6. Acceptance of study participation by the responsible project leader and commitment of online documentation of primary histopathological and clinical data as well as follow up data when assessed.

Primary outcome measures:

(1) Progression-free survival, defined as time from TMMR to a local or regional relapse, of a distant metastasis or to death of any cause whichever event comes first. Simultaneous occurrence of pelvic and distant metastases is considered as distant but should be documented in detail.

Secondary efficacy measures:

1. Overall survival, defined as time from TMMR to death of any cause; Rate of locoregional relapse and rate of distant metastases at 3 years.
2. Postoperative dysfunction of the bladder/urethra and of psychosexual function, assessed as described in the urogynecological and psychosexual subprotocol.

Secondary safety measures:

1. Therapy-induced morbidity on bladder/urethra, rectum/bowel, vagina/vulva, assessed by the LENT-SOMA scoring system at the following times after surgery: subjective scale on day 1, week 1 and 2, month 3; subjective and objective scale on month 12 and 24. The questionnaires developed by Davidson (7) will be used; Time from surgery to first micturition; Acute complications of surgery; adverse and serious adverse events.
2. Quality of life by EORTC-QLQ-C30 questionnaire at 12 and 24 months after surgery.

Aim of the study is to assess recurrence rate and morbidity following TMMR/LNE without additional radiotherapy in a multicentric observation of clinical routine treatment. In addition standardization of radical hysterectomy and of pathological work up for stage Ib to IIa cervical cancer will be achieved as described in "Requirements of participating centers". Two primary endpoints will be investigated, ranked according to their relevance: (1) PFS and (2) Late effects on bladder/urethra, measured by the subjective scale of the LENT-SOMA system. A hierarchical strategy will be used.

Further time to event endpoints will be illustrated by Kaplan-Meier plots and analyzed like the primary endpoint see above.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cervical cancer: squamous cell carcinoma or adenocarcinoma; FIGO stages IB - IIA (preoperatively); Karnofsky-Index ≥ 70; unrestricted operability; BMI <35; age >=18 years.
* Individual decision for treatment of TMMR and therapeutic LNE without adjuvant radiotherapy by the responsible clinic (clinician) on a clinical routine basis.
* Informed consent of the patient

Exclusion criteria:

* Neuroendocrine differentiation and all preoperative FIGO stage IA or >IIA;
* Distant metastases except in para-aortic lymph nodes; sclerodermia, lupus erythematodes, mixed connective tissue disease; secondary malignancy; previous radiotherapy of the pelvis.
* Patients with diseases of the connective tissue will be excluded because of unforeseeable (e.g. neurological) symptoms and disorders after surgery. Patients with a BMI ≥ 35 will be excluded because of very high risks regarding wound healing, infections and thrombosis independent on the type of surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical cancer Stages IB - IIA treated with TMMR and tLNE.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 60 months
  Progression-free survival, defined as time from TMMR to a local or regional relapse, of a distant metastasis or to death of any cause whichever event comes first. Simultaneous occurrence of pelvic and distant metastases is considered as distant but should be documented in detail.

SECONDARY OUTCOMES:
Overall Survival | 60 months
  Overall survival, defined as time from TMMR to death of any cause; Rate of locoregional relapse and rate of distant metastases at 3 years.

OTHER OUTCOMES:
Sexual and bladder function | 24 months
  Postoperative dysfunction of the bladder/urethra and of psychosexual function, assessed as described in the urogynecological and psychosexual subprotocol
Quality of Life | 60 months
  Postoperative Quality of Life as measured by the EORTC-QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Kimmig, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Hockel M, Horn LC, Hentschel B, Hockel S, Naumann G. Total mesometrial resection: high resolution nerve-sparing radical hysterectomy based on developmentally defined surgical anatomy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):791-803. doi: 10.1111/j.1525-1438.2003.13608.x. PMID 14675316
- [Background] Hockel M. Do we need a new classification for radical hysterectomy? Insights in surgical anatomy and local tumor spread from human embryology. Gynecol Oncol. 2007 Oct;107(1 Suppl 1):S106-12. doi: 10.1016/j.ygyno.2007.07.049. Epub 2007 Aug 28. PMID 17727931
- [Background] Hockel M, Horn LC, Tetsch E, Einenkel J. Pattern analysis of regional spread and therapeutic lymph node dissection in cervical cancer based on ontogenetic anatomy. Gynecol Oncol. 2012 Apr;125(1):168-74. doi: 10.1016/j.ygyno.2011.12.419. Epub 2011 Dec 8. PMID 22155677
- [Derived] Buderath P, Stukan M, Ruhwedel W, Strutas D, Feisel-Schwickardi G, Wimberger P, Kimmig R. Total mesometrial resection (TMMR) for cervical cancer FIGO IB-IIA: first results from the multicentric TMMR register study. J Gynecol Oncol. 2022 Jan;33(1):e9. doi: 10.3802/jgo.2022.33.e9. Epub 2021 Dec 6. PMID 34910390